CLINICAL TRIAL: NCT05681559
Title: Investigation of Medical Management to Prevent Episodes of Diverticulitis (IMPEDE) Trial
Brief Title: Investigation of Medical Management to Prevent Episodes of Diverticulitis Trial
Acronym: IMPEDE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, David Flum, Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00015672; 1R01DK131694-01A1 (NIH)
Record Dates: First submitted 2022-11-23; First posted 2023-01-12 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Diverticulitis
MeSH Terms: conditions — Diverticulitis | interventions — Proto-Oncogene Proteins c-raf

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medi for All (Active Comparator): Participants randomized to the USDA Mediterranean-style Food Pattern Arm (called Medi for all) will have access to a "toolbox" that includes education materials (e.g., food pattern tables according to daily caloric intake), recipes, grocery lists, group-based online dietary support, feedback, and reminders to encourage dietary change. Recipes and grocery lists can be individualized to a participant's food budget and preferences. Materials will be available in print and Web-based. This state-of-the art intervention will then use electronic feedback in the form of nudge messages designed to motivate participants to sustain or improve adherence to the Med-style Food Pattern.
  Interventions: Behavioral: Medi for All
- Fiber Supplementation (Active Comparator): Participants randomized to the High Fiber Diet Arm will be given commonly used patient education pamphlet,149 describing fiber and high-fiber foods, the rationale for increasing fiber intake, and ways patients can promote greater intake. Based on prior observational studies of incident diverticulitis, at least 25 grams/day of fiber will be recommended for participants.
  Interventions: Dietary Supplement: Standard Fiber Supplementation

INTERVENTIONS:
Behavioral: Medi for All — Please see description of Medi for All arm
  Arms: Medi for All
Dietary Supplement: Standard Fiber Supplementation — Please see description of Fiber Supplementation arm
  Arms: Fiber Supplementation

SUMMARY:
This is a randomized trial (n=75) of a Mediterranean style Food Pattern and versus standardized guidance on fiber intake for patients with diverticulitis to evaluate the feasibility of this dietary intervention including willingness to randomize and adherence to a Med-style dietary pattern. The investigators will employ state-of-the-art behavioral interventions in the form of electronic feedback to improve health-related behaviors and support dietary customization based on participants' budget, dietary preferences, and restrictions. The investigators will also examine plasma inflammatory biomarkers (interleukin-6, interleukin-10, and interleukin-1β) and fecal calprotectin at baseline, 6, and 12 months.

DETAILED DESCRIPTION:
This is a feasibility-focused, patient-level randomized trial of an intervention promoting the United States Department of Agriculture (USDA) Healthy Med-Style food pattern versus standardized guidance on fiber intake (standard educational materials related to a high-fiber diet) in patients with a history of diverticulitis. This trial will assess and address barriers to the eventual large-scale trial and lay groundwork for that trial that will focus on the risk of recurrent diverticulitis and other clinical outcomes. The investigators will also compare changes in serum and stool biomarkers of inflammation that are proximal endpoints in the causal path relating a Mediterranean diet pattern's anti-inflammatory properties and recurrence of diverticulitis.

Participants randomized to the USDA Mediterranean-style Food Pattern Arm (called Medi for all) will have access to a "toolbox" that includes education materials (e.g., food pattern tables according to daily caloric intake), recipes, grocery lists, group-based online dietary support, feedback, and reminders to encourage dietary change. Recipes and grocery lists can be individualized to a participant's food budget and preferences. Materials will be available in print and Web-based. This state-of-the art intervention will then use electronic feedback in the form of nudge messages designed to motivate participants to sustain or improve adherence to the Med-style Food Pattern. Every two weeks, participants in the intervention arm will be prompted via a digital online platform (analog also available) to complete the 14-item Mediterranean Diet Assessment Score (MEDAS) (an adapted version of the MEDAS Score previously used in the Prevencion con Dieta Mediterranea [PREDIMED study]) for the purpose of providing timely, individual feedback on diet adherence (not for assessing adherence to the diet pattern). The MEDAS score will be calculated via the online digital platform and ranked according to 3 cutpoints: ≤7, 8-9, or ≥10. Patients will be encouraged to achieve a score of ≥10 which is considered high adherence. The platform will then offer feedback based on the levels of self-reported adherence to the diet including self vs. peer comparisons and support resources. Nudge messages will utilize information from a baseline assessment of participants' dietary attitudes and beliefs about which food groups within a Med-style food pattern they perceive to be most within their control. Ultimately, this approach will enable us to provide participants with dietary information and services that support adherence by accounting for attitudes, norms, and perceived control. The extent of interaction with the online platform will be assessed bi-weekly; degree of adherence to the USDA Med-style food pattern; and engagement in dietician services will be assessed at quarterly intervals.

Participants randomized to the High Fiber Diet Arm will be given commonly used patient education pamphlet, describing fiber and high-fiber foods, the rationale for increasing fiber intake, and ways patients can promote greater intake. Based on prior observational studies of incident diverticulitis, at least 25 grams/day of fiber will be recommended for participants.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥18 years;
* Patients presenting (or recently presented) to gastroenterologist or surgeons or accessing study website after recovery from an episode of diverticulitis (within the prior 18 months), either the index episode or recurrent.
* Ability to provide written informed consent in English.

Exclusion Criteria:

* Unable or unwilling to return for specimen collection visits or be contacted for and/or complete research surveys;
* Currently incarcerated in a detention facility or in police custody (patients wearing a monitoring device can be enrolled) at baseline/screening;
* Last episode of acute diverticulitis currently unresolved (i.e., on antibiotics for diverticulitis; drain in place);
* Intolerance/allergy to the main components of the Med-style food pattern;
* Surgery for diverticulitis within past 6 months without an episode of diverticulitis post-surgery;
* Planned elective surgery in next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Willingness to enroll | through study completion, over a period of 2 years
  Number of randomized participants out of number approached
Adherence to Med-Style Food Pattern | through study completion, over a period of 12 months
  Med-style Pattern score calculated from the Nutrition Assessment Shared Resource Food Frequency Questionnaire
Participant retention | through study completion, over a period of 12 months
  Proportion enrolled and retained at 3, 6, 9 and 12 months
Engagement with nutrition services | Quarterly through study completion, over a period of 12 months
  Number of sessions with dietician
Interaction with online program | Bi-weekly through study completion, over a period of 12 months
  Number of times accessed

SECONDARY OUTCOMES:
Change in Plasma, Interleukin (IL)-6, IL-10, IL-1b, fecal calprotectin | Baseline, 6, 12 months through study completion, over a period of 12 months
  Concentration
Diverticulitis events | Quarterly through study completion, over a period of 12 months
  Self-reported (presumed), subset of those resulting in healthcare utilization (e.g., hospitalization, surgery).
National Surgical Quality Improvement Program (NSQIP)-defined complications, a subset of which are serious adverse events to be reported to Independent Safety Monitor | Quarterly through study completion, over a period of 12 months
  Standardized assessment-serious events defined as death, cardiac arrest, myocardial infarction, pneumonia, progressive renal insufficiency, acute renal failure, pulmonary embolism, deep vein thrombosis, return to operating room, serious site infections
Change in Diverticulitis Quality of Life Survey (DVQOL) | Baseline, 6, 12 months
  A 17-item questionnaire that assesses four domains: symptoms, concerns, emotions, and behavior changes related to diverticulitis, ranging from 0 (best) to 10 (worst)
Change in Gastrointestinal Quality of Life Index (GIQLI) | Baseline, 6, 12 months
  A 36-item questionnaire that assesses five domains: gastrointestinal symptoms, physical function, emotional well-being, social well-being, and perception of medical treatment measured by a single item question. Each item has 5 response choices (i.e., all of the time, most of the time, some of the time, a little of the time, never). In addition, the measure produces an overall QoL score (0-144) where higher numbers indicate greater QoL.
Change in International Physical Activity Questionnaire (IPAQ) short form | Baseline, 6, 12 months
  A validated 7-item questionnaire: moderate and vigorous physical activity, walking, and sitting in the past 7 days. Output is self-reported minutes of moderate and vigorous physical activity as well as walking from which weekly moderate and vigorous physical activity, sitting, and walking can be assessed.
Healthcare utilization | Quarterly through study completion, at 3, 6, 9, 12 months
  Counts of ED/hospital encounters, diverticulitis-related diagnostic/therapeutic interventions
Change in self-reported weight | Baseline, 6, 12 months
  Self-reported weight

CONTACTS AND LOCATIONS:
Overall Officials: David R Flum, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/59/NCT05681559/Prot_SAP_001.pdf